CLINICAL TRIAL: NCT06583343
Title: Evaluation of the Effect of Botulinum Toxin Application on Selective Motor Control and Pain in Children Diagnosed With Diplegic Cerebral Palsy
Brief Title: Effect of Botulinum Toxin on Selective Motor Control and Pain in Diplegic Cerebral Palsy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREH-FTR-OB-01
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy Spastic Diplegia
Keywords: Cerebral Palsy; Selective Motor Control; Botulinum Neurotoxin Injection; Spasticity; Pain
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: One group receiving conventional physical therapy as the control group, along with another experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Conventional Physical Therapy Group (Active Comparator): Conventional rehabilitation, personalized and administered under the guidance of a physiotherapist
  Interventions: Other: Conventional Physical Therapy
- Botulinum toxin injection group (Active Comparator): Administration of botulinum toxin injection prior to the conventional rehabilitation program
  Interventions: Drug: OnabotulinumtoxinA; Other: Conventional Physical Therapy

INTERVENTIONS:
Drug: OnabotulinumtoxinA — Botulinum toxin injections were administered in appropriate doses to the spastic muscles of children with cerebral palsy.
  Other Names: botox
  Arms: Botulinum toxin injection group
Other: Conventional Physical Therapy — Conventional rehabilitation program; consisting of walking-balance exercises, range of motion exercises, stretching, and strengthening exercises, was provided for 1 hour, 5 days a week, totaling 30 sessions

SUMMARY:
The aim of this study is to investigate the effects of Botulinum Neurotoxin-A (BoNT-A) injection applied to spastic muscles on pain sensation and Selective Motor Control (SMC) in cases diagnosed with diplegic spastic Cerebral Palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a non-progressive, permanent neurological disorder that occurs in the fetal or infant brain. CP, defined as a group of non-progressive movement and posture disorders, is the most common cause of neurological disability in children. The primary cause is insufficient oxygen supply to the fetus and brain asphyxia. However, other underlying factors may also be involved. Preterm birth is the most important risk factor that should be considered first.

Musculoskeletal problems mainly arise due to positive findings such as spasticity, clonus, hyperreflexia related to Upper Motor Neuron damage, and negative findings such as weakness and reduced Selective Motor Control (SMC).

Selective Motor Control (SMC) is the ability to achieve muscle activation in an appropriate pattern, in an isolated manner, to produce a voluntary movement or posture. Studies have shown that the impact of SMC on motor performance is as significant as routinely measured issues such as spasticity and contracture.

Pain is a common problem in CP, with more than half of children and adults with CP reporting pain as an issue. Assessing pain in children with CP is particularly challenging, especially in those who cannot express themselves verbally. The most common potential causes of pain include neuromuscular problems such as muscle spasms, musculoskeletal problems like hip dislocation and scoliosis, and gastrointestinal issues such as gastroesophageal reflux and constipation.

Botulinum Neurotoxin-A (BoNT-A), when applied intramuscularly, inhibits presynaptic acetylcholine (Ach) release by preventing the fusion of Ach vesicles with the plasma membrane. BoNT-A acts on the motor endplate, providing reversible chemical denervation. It is used for localized spasticity and can be applied to multiple muscles in a single session. It is generally used for spasticity starting from the age of 2. Along with rehabilitation, it aids in motor learning, promotes functional progression, and delays or prevents the development of orthopedic deformities.

The aim of our study is to investigate the effects of BoNT-A injections into spastic muscles on pain perception and SMC in patients with diplegic spastic CP.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Cerebral Palsy
* Between the ages of 4-12
* GMFCS (Gross Motor Function Classification System)1-4
* Patients who have received an appropriate indication for BoNT-A injection from an experienced physiatrist
* Patients who have not had botulinum toxin administered in the last 6 months

Exclusion Criteria:

* Mental retardation
* GMFCS 5
* Have an intrathecal baclofen pump for spasticity treatment or history of soft tissue and/or bone surgery
* Underwent dorsal rhizotomy
* Have an active infection or a localized skin infection at the injection site
* Using aminoglycoside antibiotics
* Contracture

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
SCALE (Selective Control Assessment of the Lower Extremity) | six weeks
  SCALE; it is a scale that can be easily applied in outpatient clinic conditions, does not require any equipment. A total of 5 regions are assessed: the hip, knee, ankle, subtalar joint, and toes.
  Scoring is as follows: 0 (cannot be performed), 1 (impaired SMC), and 2 (normal). If the patient performs the movement correctly within 3 seconds, without moving any other joint besides the one being evaluated and without any mirror movement, it is considered normal SMC (2 points). If there is movement in another joint, mirror movement occurs, the range of motion is less than 50% of the passive ROM (Range Of Motion), or the movement takes longer than 3 seconds, it is considered impaired SMC (1 point). If the patient cannot initiate the movement or develops flexor/extensor synergy, it is scored as unachievable (0 points).
Boyd and Graham SMC Test | six weeks
  This test, developed by Boyd and Graham, aims to evaluate the Selective Motor Control (SMC) of ankle dorsiflexion. The test assesses the patient's ability to activate the muscles responsible for ankle dorsiflexion (DF). It consists of 5 items and is scored on a scale from 0 to 4.
  0: No movement at all when asked to dorsiflexion the foot.
  1. Limited dorsiflexion achieved primarily through the use of extensor hallucis longus (EHL) and/or extensor digitorum brevis (EDB).
  2. Limited dorsiflexion achieved using EHL, EDB, and some tibialis anterior (TA) muscle.
  3. Dorsiflexion primarily using TA, but with accompanying hip and knee flexion.
  4. Isolated selective ankle dorsiflexion (DF) achieved through isolated TA muscle activity without hip or knee flexion.
Visual Analog Scale (VAS) | six weeks
  The Visual Analog Scale (VAS) is a very simple and easy-to-use pain scale where patients assess the intensity of their pain between "no pain" (0 points) and "unbearable pain" (10 points). The patient rates their pain on a scale from 0 to 10:
  0: No pain 1-3: Mild pain 4-6: Moderate pain 7-10: Severe pain

SECONDARY OUTCOMES:
SCUES (Selective Control of the Upper Extremity Scale) | six weeks
  SCUES; is a test that does not require special equipment and can be completed in less than 15 minutes. It evaluates a total of 5 joints in relation to their fundamental movement patterns: shoulder (abduction/adduction), elbow (flexion/extension), forearm (supination/pronation), wrist (flexion/extension), and fingers (grasp/release). Each joint is scored on a four-point scale:
  0: No SMC (Selective Motor Control)
  1. Moderately reduced SMC
  2. Slightly reduced SMC
  3. Normal SMC
  The patient is seated, and the evaluator first demonstrates the appropriate movement on themselves. Then, the evaluator demonstrates the movement passively on the patient and asks the patient to replicate the movement. Four key indicators of impaired SMC are:
  1. Presence of mirror movements
  2. Movement of joints other than the target joint
  3. Presence of trunk movements
  4. Inability to achieve passive end-range of motion during dynamic movement
Functional Independence Measure for Children (WeeFIM) | six weeks
  It evaluates the effects of developmental problems on independence at home, school, and in the community. It guides clinicians in determining the level of daily living activities and motor skills in patients with CP, protecting them from potential secondary problems, predicting prognosis, and assessing the need for assistive devices.
Pediatric Quality of Life Inventory (PedsQL) | six weeks
  It is designed to assess the quality of life in children and adolescents aged 2-18 years. There are a total of 4 subscales evaluating physical, emotional, social, and school-related functioning, with a total of 23 items. Each item is scored based on the response as 100, 75, 50, 25, or 0, then summed, and the total score is divided by the number of items to obtain the score for the corresponding subscale.
Child and Adolescent Participation Questionnaire (CASP) | six weeks
  The CASP is a questionnaire that assesses the participation of patients with CP in various environments (such as home, school, and neighborhood). It consists of 4 subscales and 20 questions. Each item is scored on a scale from 0 to 4. As the total score increases, the individual's level of participation increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Yılmaz Yalçınkaya, Principal Investigator — Gaziosmanpasa Research and Education Hospital; Ozan Baş, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No